CLINICAL TRIAL: NCT02547870
Title: A Phase 1 Open-Label, Randomized, Parallel-Group Study in Healthy Subjects to Investigate the Effect of Different Storage Conditions of a Long-Acting Nanosuspension of Rilpivirine on the Single-Dose Plasma Pharmacokinetics of Rilpivirine After Intramuscular Injection
Brief Title: A Study to Evaluate the Pharmacokinetic Effects of Different Storage Conditions for a Long-Acting Nanosuspension of Rilpivirine on Pharmacokinetics
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Infectious Diseases BVBA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR107976; TMC278LAHTX1001 (Other: Janssen Infectious Diseases BVBA); 2015-002259-92 (EudraCT Number)
Record Dates: First submitted 2015-09-10; First posted 2015-09-11 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Human Immunodeficiency Virus Type 1
Keywords: Rilpivirine; Healthy participants
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

ARMS (2):
- Rilpivirine Long-Acting Parenteral Formulation (RPV-LA) (Experimental): Participants will receive oral tablet of rilpivirine 25 milligram (mg) once on Day 1 of session 1 and intramuscular (IM) injection of rilpivirine long-acting parenteral formulation 600 mg once on day 1 of session 2.
  Interventions: Drug: Rilpivirine (RPV); Drug: Rilpivirine Long-Acting Parenteral Formulation (RPV-LA)
- Aged RPV-LA (Experimental): Participants will receive oral tablet of rilpivirine 25 milligram (mg) once on Day 1 of session 1 and IM injection of aged rilpivirine long-acting parenteral formulation 600 mg once on day 1 of session 2.
  Interventions: Drug: Rilpivirine (RPV); Drug: Aged RPV-LA

INTERVENTIONS:
Drug: Rilpivirine (RPV) — Participants will receive one oral tablet of rilpivirine 25 milligram (mg) once on Day 1 of session 1.
Drug: Rilpivirine Long-Acting Parenteral Formulation (RPV-LA) — Participants will receive one intramuscular (IM) injection of rilpivirine long-acting parenteral formulation 600 mg once on day 1 of session 2.
  Arms: Rilpivirine Long-Acting Parenteral Formulation (RPV-LA)
Drug: Aged RPV-LA — Participants will receive one intramuscular (IM) injection of aged rilpivirine long-acting parenteral formulation 600 mg once on day 1 of session 2.
  Arms: Aged RPV-LA

SUMMARY:
The purpose of this study is to compare the single-dose pharmacokinetics of rilpivirine (RPV) after intramuscular (IM) injection of rilpivirine long-acting parenteral formulation (RPV-LA) and 'aged' RPV-LA, in healthy adult participants.

DETAILED DESCRIPTION:
This is a phase 1 randomized (study medication is assigned by chance), open-label (all people know the identity of the intervention), parallel-group, sequential study in healthy adult participants to investigate the effect of different storage conditions for RPV-LA on the single-dose pharmacokinetics of rilpivirine (RPV) after intramuscular injection. A total of 60 healthy adult participants will be enrolled in this study. The study will consist of 2 treatment sessions in a fixed sequential order : session 1 of up to day 8, all participants will receive a single oral dose of rilpivirine 25 milligram (mg) tablet on day 1, session 2 will consists of 2 treatment groups. The participants will be randomized in session 2 on Day 1 in a 1:1 ratio to Treatments A and B. Each treatment group will receive one IM injection of RPV LA on Day 1 of session 2. Session 1 and 2 will be separated by a washout period of at least 14 days. The total study duration for each participant will be approximately 6.5 months. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Each participant must sign an Informed Consent Form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and are willing to participate in the study
* Participant must be willing and able to adhere to the prohibitions and restrictions specified in this protocol
* Participant must be healthy on the basis of a medical evaluation that reveals the absence of any clinically significant abnormality and includes a physical examination, medical history, vital signs, Electrocardiogram (ECG), and the results of blood biochemistry, hematology and coagulation tests and a urinalysis performed at Screening
* A female participant of childbearing potential must have a negative serum (beta-human chorionic gonadotropin [beta-hCG]) at Screening and a negative urine pregnancy test on day 1
* Participant must be non-smoking for at least 3 months prior to selection

Exclusion Criteria:

* Female participant who is breastfeeding at Screening
* Participants with a history of any illness that, in the opinion of the investigator, might confound the results of the study or pose an additional risk in administering study drug to the participant or that could prevent, limit or confound the protocol specified assessments. This may include, but is not limited to, renal dysfunction, significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic, rheumatologic, psychiatric, neoplastic, or metabolic disturbances
* Has known allergies, hypersensitivity, or intolerance to rilpivirine (RPV) or its excipients
* Has a history of drug allergy such as, but not limited to, sulfonamides and penicillins, or drug allergy witnessed in previous studies with experimental drugs
* Having donated or lost more than 1 unit of blood (500 milliliter [mL]) within 60 days or more than 1 unit of plasma within 7 days before the first dose of study drug

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2015-08-14 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2016-04-26 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  The Cmax is the maximum observed plasma concentration of rilpivirine.
Area Under the Plasma Concentration-Time Curve From Time Zero (Day 1) to Day 28 (AUC[0-d28]) | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120 and 168 hours post-dose
  The AUC (0-d28) is the area under the plasma concentration-time curve for rilpivirine from time zero to day 28.
Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Time (AUC [0-last]) | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  The AUC (0-last) is the area under the plasma concentration-time curve for rilpivirine from time zero to last quantifiable time.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z); wherein AUC(last) is area under the plasma concentrationtime curve from time zero to last quantifiable time, C(last) is the last observed quantifiable concentration, and lambda(z) is elimination rate constant.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events | Up to 180 Days
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Time to reach the maximum observed plasma concentration (Tmax) | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  The Tmax is the actual sampling time to reach maximum observed plasma concentration of rilpivirine.
Elimination Rate Constant (Lambda [z]) of rilpivirine | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  The Lambda (z) determined by linear regression of the terminal points of the ln-linear plasma concentration-time curve.
Apparent Terminal Half-life (t[1/2]) of rilpivirine | In session1: Pre-dose, 0.5, 1, 2, 3, 4, 5, 6, 9, 12, 16, 24, 48, 72, 120 and 168 hours post-dose; In session 2: Pre-dose, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168,216, 264, 336, 408, 528, 672, 1344, 2016, 2688, 3360 and 4032 hours post-dose
  Apparent terminal elimination half-life, calculated as 0.693/Lambda (z).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Infectious Diseases BVBA Clinical Trial, Study Director — Janssen Infectious Diseases BVBA
Locations (1):
- Antwerp, Belgium